CLINICAL TRIAL: NCT03547544
Title: Effectiveness of Rapid Urease Test (Helicotec) for The Diagnosis of Helicobacter Pylori Infection in Dyspepsia Patients in Endoscopy Centre
Brief Title: Rapid Urease Test for Diagnosis Helicobacter Pylori Infection
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Staff of Gastroenterology Division, Internal Medicine Department, Indonesia University
Other Study IDs: 18-04-0394
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori; urease test; helicotec

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, the gold standard examinations for diagnosing H. pylori infection are histopathology and culture examination. However, those examinations take long preparation so they are not suitable to be applied in daily practice. In progress, another examination is being developed to detect urease enzyme from tissue biopsy. It is relatively faster in diagnosing H. Pylori infection. Some commercial urease tests which are available in Indonesia are Helicotec® and Pronto Dry®.

This study aims to determine the effectivity of Helicotec® in diagnosing H. pylori infection. It is expected to be scientific evidence that can be used as the basis daily routine of urease test in diagnosing H. Pylori infection.

DETAILED DESCRIPTION:
This study is a diagnostic study. There will be 97 dyspepsia patients who met the inclusion and exclusion criteria. They will answer the questionnaire about personal data and examined physically. They will also undergo endoscopy, biopsy, and urease test using Helicotec®

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-55 years old),
* Diagnosed with dyspepsia,
* Indicated for endoscopy,
* Agreed to participate in the study and signed the informed consent.

Exclusion Criteria:

* Pregnancy and breastfeeding woman,
* Patients with alarm symptom,
* History taking of antibiotics (amoxicillin, clarithromycin, levofloxacin), H2 receptor antagonist, proton pump inhibitor, misoprostol, sucralfat, bismuth, NSAIDs, steroid, rheumatoid drug within the last 2 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: General population: Jakarta citizen Targeted population: Patients of endoscopy centre Cipto Mangunkusumo Hospital Sample: Targeted population who undergo endoscopy examination and met the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Effectivity of Helicotec | 1 day
  Obtained the sensitivity and specificity value

CONTACTS AND LOCATIONS:
Overall Officials: Ari F Syam, Dr, MD, Principal Investigator — Gastroenterology Division, Internal Medicine Department RSCM/UI
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No